CLINICAL TRIAL: NCT06762223
Title: Intervention of Henagliflozin on Liver Fibrosis in Patients with Metabolic Dysfunction Associated Steatotic Liver Disease (MASLD) and Type 2 Diabetes Mellitus (T2DM)
Brief Title: Henagliflozin on Liver Fibrosis in Patients with MASLD and T2DM
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xiqiao Zhou (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Xiqiao Zhou, Professor, Jiangsu Province Hospital of Traditional Chinese Medicine
Organization: Jiangsu Province Hospital of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024NL-195-01
Record Dates: First submitted 2024-12-17; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Metabolic Dysfunction-associated Steatotic Liver Disease; Type 2 Diabetes Mellitus
Keywords: metabolic dysfunction-associated steatotic liver disease; type 2 diabetes mellitus; Henagliflozin; SGLT2i; Liver fibrosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Liver Cirrhosis | interventions — henagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: In the process of randomizing groups, the study designers assigned a blinded code to each participant. This coding is organized based on the order of enrollment.Only the study implementer will have access to the serial numbers of the study subjects, the blinded codes, and the drugs labeled with those codes. The details of the blind codes are known solely to the lead study designers and are maintained by designated personnel. At this stage, as the study implementer includes participants in sequence, only the drugs labeled with the corresponding codes can be administered, ensuring that neither the implementer nor the participants are aware of the group assignments or the drugs being used.To assess the quality of blinding completion, we employed the James Blinding Index (JBI) and the Bang Blinding Index (BBI) as evaluative tools.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Control Group (Placebo Comparator): Placebo + Metformin 1.7g/d
  Interventions: Drug: Metformin 1700 mg daily; Other: Placebo of Henagliflozin
- Intervention Group (Experimental): Henagliflozin 10mg/d + Metformin 1.7g/d
  Interventions: Drug: Henagliflozin 10 mg daily; Drug: Metformin 1700 mg daily

INTERVENTIONS:
Drug: Henagliflozin 10 mg daily — Henagliflozin (SHR3824) is a hypoglycemic agent classified as an SGLT2i, which has been independently developed by Jiangsu Hengrui Pharmaceutical Co., Ltd. (China) and Shanghai Hengrui Pharmaceutical Co., Ltd (China). It received marketing authorization in China on December 31, 2021 (ID: H20210053).The prescribed dosage of Henagliflozin is 10 mg per day, as indicated on the drug label, with administration recommended in the early morning. In instances where a participant forgot to take the medication in the morning, they were permitted to do so until 12:00 PM on the same day.
  Arms: Intervention Group
Drug: Metformin 1700 mg daily — The metformin utilized in this study is Metformin Hydrochloride Extended-release Tablets, manufactured by Bristol-Myers Squibb Company. This formulation of metformin is available in a dosage of 0.85 grams per tablet, necessitating that patients administer two tablets daily to acquire the dose of 1.7g daily, to be taken within thirty minutes prior to breakfast and dinner respectively. However, adjustments to the metformin dosage were not permitted during follow-up visits.
Other: Placebo of Henagliflozin — The placebo was supplied by the pharmaceutical company responsible for Henagliflozin, ensuring that both the placebo and Henagliflozin were indistinguishable in terms of appearance, taste, and odor, while lacking any significant pharmacological effect. Administration of the placebo was recommended to occur in the early morning.
  Arms: Control Group

SUMMARY:
The prevalence of metabolic dysfunction-associated steatotic liver disease (MASLD) is increasing due to changes in economic conditions and lifestyle, and it is anticipated to become a significant liver disease burden in the future. This is particularly true for patients with MASLD who also have type 2 diabetes mellitus (T2DM), as the rate of comorbidity between these conditions has risen in recent years due to their shared mechanisms, necessitating careful management of both. Liver fibrosis is a critical concern, as poor blood glucose control can worsen liver fibrosis, which in turn complicates blood sugar management. Therefore, addressing liver fibrosis in patients with MASLD and T2DM is urgent, yet there are currently no targeted therapies to reverse its progression. SGLT2 inhibitors, have shown promise in potentially reversing liver fibrosis, but existing research is limited and has not adequately focused on liver fibrosis improvement, highlighting the need for more robust evidence-based studies.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be aged between 18 and 75 years.
2. Participants must meet the diagnostic criteria for MASLD and T2DM.
3. Participants' HbA1c level between 6.5% and 9%.
4. The LSM obtained via the FibroScan device must be equal to or greater than 8 kPa.
5. Participants must not have experienced a significant change in body weight exceeding 15% within the past four weeks.
6. Participants must not have utilized non-biguanide hypoglycemic medications in the three months preceding the study.

Exclusion Criteria:

1. Patients diagnosed with non-MASLD, which encompasses conditions such as viral hepatitis, autoimmune liver disease, liver tumors, and drug-induced liver injury, among others;
2. Individuals exhibiting ALT and/or AST levels that exceed the normal range by threefold or more;
3. Patients currently using or having used medications associated with secondary MASLD (including, but not limited to, corticosteroids, estrogen, amiodarone, methotrexate, etc.) within the preceding three months;
4. Individuals utilizing or having utilized medications within the last three months that possess the potential to ameliorate hepatic steatosis or fibrosis in MASLD (including, but not limited to, ursodeoxycholic acid, bicyclol tablets, silymarin capsules, polyene phosphatidylcholine capsules, vitamin E, etc.);
5. Patients with known or suspected elevated alcohol consumption (females exceeding 12 grams per day; males exceeding 24 grams per day) or those on medications that may contribute to increased consumption;
6. Individuals who have experienced severe acute complications such as hypoglycemia, ketoacidosis, hyperglycemia, or hyperosmolar states within the past month or during the course of medication;
7. Patients who have undergone metabolic bariatric surgery or are currently participating in bariatric treatment;
8. Individuals with significant primary systemic pathologies, including but not limited to respiratory, circulatory, digestive, urinary, neurological, hematological, rheumatological, endocrine diseases, tumors, or AIDS;
9. Female participants who are pregnant, breastfeeding, or of childbearing potential and not employing a highly effective contraceptive method;
10. Individuals with known allergies or potential allergies to the medications utilized in this study, rendering them intolerant;
11. Patients with a history of recurrent or severe urinary and genital tract infections;
12. Individuals exhibiting severe cognitive impairment or mental illness that impedes their ability to cooperate;
13. Patients currently engaged in clinical observation of other pharmacological agents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Liver stiffness measurements (LSM) of subjects | From enrollment to the treatment at 24 and 48 weeks
  As determined by magnetic resonance elastography (MRE)

SECONDARY OUTCOMES:
Efficacy Evaluation of MASLD in fibrosis | From enrollment to the treatment at 24 and 48 weeks
  This includes:
  1. Difference from baseline in LSM of subjects based on FibroScan;
  2. The proportion of LSM of subjects on MRE reduced by ≥15%;
  3. The proportion of LSM of subjects on FibroScan reduced by ≥15%
Efficacy Evaluation of MASLD in liver fatty quantification | From enrollment to the treatment at 24 and 48 weeks
  This includes:
  1. Difference from baseline in liver fatty quantification of subjects based on magnetic resonance imaging proton density fat fraction(MRI-PDFF);
  2. Difference from baseline in liver fatty quantification of subjects based on FibroScan;
  3. The proportion of liver fatty quantification of subjects based on MRI-PDFF was reduced by ≥30%;
  4. The proportion of liver fatty quantification of subjects based on FibroScan was reduced by ≥30%;
Efficacy Evaluation of MASLD in non-invasive biological indicators related to liver fibrosis | From enrollment to the treatment at 24 and 48 weeks
  This includes:1.NAFLD fibrosis score(NFS) = - 1.675 + [0.037 ×Age] + [0.094 × body mass index(BMI) (kg/m2)] + [1.13 × fasting plasma glucose(FPG)/ Diabetes (Yes=1，No= 0)] + [0.99 × aspartate aminotransferase(AST)/alanine aminotransferase(ALT)] - [0.013 × platelet count(PLT) (×109/L)] - [0.66 × Albumin(ALB) (g/dL)]; NFS <-1.455, -1.455-0.675, and >0.675 mean expressed as low, medium, and high risk, respectively(39); 2.Fibrosis-4(FIB-4) index= [Age× AST (U/L)]/[PLT (×109/L)× ALT (U/L)1/2];
Renal function | From enrollment to the treatment at 24 and 48 weeks
  This includes:This includes:Difference from baseline in renal function related parameters of subjects, primarily including uric acid(UA), urea nitrogen(BUN), creatinine(Cr), urine albumin-to-creatinine ratio(UACR).
Liver function | From enrollment to the treatment at 24 and 48 weeks
  This includes:Difference from baseline in liver function related parameters of subjects, primarily including AST, ALT, gamma-glutamyl transferase(GGT), alkaline phosphatase(ALP), ALB, total bilirubin(TBiL).
Lipid metabolism | From enrollment to the treatment at 24 and 48 weeks
  This includes:Difference from baseline in lipid metabolism related parameters of subjects, primarily including Triglyceride(TG), total cholesterol(TC), low-density lipoprotein cholesterol(LDL-C), high-density lipoprotein cholesterol(HDL-C).
Efficacy Evaluation of T2DM | From enrollment to the treatment at 24 and 48 weeks
  FPG
Efficacy Evaluation of T2DM | From enrollment to the treatment at 24 and 48 weeks
  fasting insulin concentrations(FINS)
Efficacy Evaluation of T2DM | From enrollment to the treatment at 24 and 48 weeks
  fasting C-peptide(FCP)
Efficacy Evaluation of T2DM | From enrollment to the treatment at 24 and 48 weeks
  hemoglobin A1c(HbA1c)
Efficacy Evaluation of T2DM | From enrollment to the treatment at 24 and 48 weeks
  homeostatic model assessment of insulin resistance(HOMA-IR)

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu province hospital of traditional chinese medicine, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No